CLINICAL TRIAL: NCT01188291
Title: Retinal Nerve Fiber Layer Thickness Measurements Using Optical Coherence Tomography in Patients With Sleep Apnea Syndrome
Brief Title: Retinal Nerve Fiber Layer Thickness Measurements in Patients With Sleep Apnea Syndrome
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, Professor, Carmel Medical Center
Other Study IDs: CMC070029CTIL
Record Dates: First submitted 2010-08-17; First posted 2010-08-25 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2010-08

CONDITIONS: Obstructive Sleep Apnea; Hypopnea Syndrome; Glaucoma
Keywords: Optical Coherence Tomography; Retinal Nerve Fiber Layer Thickness; Obstructive Sleep Apnea; Hypopnea syndrome; Glaucoma
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleep Apnea / Hypopnea syndrome: Study group composed of patients with Obstructive Sleep Apnea / Hypopnea syndrome

SUMMARY:
The purpose of this study was to measure the retinal nerve fiber layer (RNFL) thickness in eyes of Obstructive Sleep Apnea/hypopnea syndrome (OSAHS) using optical coherence tomography (OCT), and assess whether it is decreased. The investigators then compared the results with healthy subjects database of RNFL thickness from another retrospective study.

DETAILED DESCRIPTION:
An association between glaucoma and OSAHS has been reported in several studies. Glaucoma is a progressive optic neuropathy involving loss of retinal ganglion cells and their axons at the level of the optic nerve head.Computerized technologies have now been successfully used in evaluating retinal nerve fiber layer (RNFL) thickness in glaucoma.Given the evidence of a possible link between OSAHS and glaucoma, it is reasonable that structural losses in retinal nerve fiber layer (RNFL) thickness would be present in OSAHS.Indeed,decreased retinal nerve fiber layers was found in patients with OSAHS, the severity of which correlated with the severity of the patients' OSAHS using scanning laser Polarimetry (SLP).Optical coherence tomography (OCT) provides quantitative RNFL thickness data by measuring the difference in the temporal delay of back-scattered light from the RNFL and a reference mirror.During the past decade, OCT has been used widely in clinical practice to discriminate glaucomatous eyes and eyes with early perimetric glaucoma from normal eyes. Several studies confirmed the accuracy and reproducibility of the RNFL thickness measurements by OCT. The thickness of the peripapillary RNFL was measured with the Stratus OCT(Carl Zeiss Meditec, Inc, Dublin,CA)using the fast scan protocol(3.4).Only good quality images, as judged by the well-focused and centered scans,no artifacts showing distorted anatomy, no missing parts and a signal strength ≥6, were used for further analysis. The considered OCT parameters were overall average RNFL thickness and the average RNFL thickness in 4 quadrants (superior, nasal,inferior,and temporal)extracted from the standard RNFL thickness analysis report(RNFL Thickness Average Analysis Protocol).

ELIGIBILITY:
Inclusion Criteria:

* formal diagnosis of moderate or severe OSAHS
* eligibility to sign informed consent form
* older than 18 years

Exclusion Criteria:

* known glaucoma
* not eligible to sign informed consent form
* younger than 18 years
* incompetent persons who lack decision making capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group composed of patients with Obstructive Sleep Apnea / Hypopnea syndrome.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer Thickness as measured Optical Coherence Tomography, and expressed in micrometers. | four months

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, Prof, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Sagiv O, Fishelson-Arev T, Buckman G, Mathalone N, Wolfson J, Segev E, Peled R, Lavi I, Geyer O. Retinal nerve fibre layer thickness measurements by optical coherence tomography in patients with sleep apnoea syndrome. Clin Exp Ophthalmol. 2014 Mar;42(2):132-8. doi: 10.1111/ceo.12145. Epub 2013 Jul 15. PMID 23777553